CLINICAL TRIAL: NCT07289061
Title: Application of Positive Psychology Interventions in Individuals With Early-stage Cognitive Decline Related to Dementia: Their Impact on Cognitive and Brain Functioning
Brief Title: Positive Psychology for Early Cognitive Decline: Effects on Cognitive and Brain Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Alzheimer Hellas (Unknown)
Responsible Party: Principal Investigator, Dimitra Vasileiou, PhD Candidate, Department of Psychology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99/5-6-2024
Record Dates: First submitted 2025-11-16; First posted 2025-12-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Subjective Cognitive Decline (SCD); Mild Cognitive Impairment (MCI); Alzheimer Dementia (AD)
Keywords: positive psychology; non-pharmacological intervention for dementia; character strengths; mindfulness; forgiveness; gratitude; humor; alzheimer's disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Parallel, two-arm randomized clinical trial. Participants with SCD or MCI are randomized within diagnosis to one of two arms: (1) multi-component Positive Psychology program delivered online (weekly small-group sessions for ~16 weeks plus brief home practice), or (2) treatment as usual (continuation of usual care with no additional structured program from the study team). Outcomes are assessed at baseline, mid-program, post-program, and follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology Intervention (Experimental): Multi-component Positive Psychology Intervention delivered online in small groups. One session per week (~60 minutes) for about 16 weeks plus brief daily home practice (about 10 minutes). Core components include identifying and using character strengths and mindfulness. Facilitated by trained psychologist. No medicines are given.
  Interventions: Behavioral: Positive Psychology Intervention
- Treatment as Usual (Active Comparator): Participants continue the treatment they already receive (e.g. cognitive training) from their usual providers. No additional structured positive psychology program is delivered by the study team. Assessments occur at the same time points as the experimental arm (baseline, mid-program, post-program, and follow-up).
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Positive Psychology Intervention — Online, group-based Positive Psychology intervention delivered by trained psychologist. One 60-minute session per week for ~16 weeks plus brief daily home practice (~10 minutes). Core components: identification and use of character strengths and mindfulness practices. Includes goal setting and habit formation. Materials provided in Greek. The sessions will take place via secure videoconference. No medications are administered. Participants will continue to receive TAU but they will have one extra hour per week for Positive Psychology Intervention.
  Arms: Positive Psychology Intervention
Behavioral: Treatment as usual (TAU) — Structured cognitive training program targeting attention, memory, and executive functions. Participants will continue to receive cognitive training at Alzheimer Hellas. Activities include paper-and-pencil and computerized tasks (e.g., working-memory, processing speed, problem solving). No Positive Psychology components are included.
  Arms: Treatment as Usual

SUMMARY:
This randomized study tests whether a new multicomponent Positive Psychology program can improve cognition and wellbeing in older adults at the earliest stages of dementia-related decline.

About 128 participants with Subjective Cognitive Decline or Mild Cognitive Impairment will be enrolled. Half will be randomized to the Positive Psychology program and half to Treatment As Usual (TAU).

The program consists of weekly, small-group online sessions for ~24 weeks plus brief home practices. All participants (both arms) will complete questionnaires and cognitive tests at baseline, during treatment, post-treatment, and 9-month follow-up.

Primary question: Do participants receiving the Positive Psychology program show better cognitive and brain-function outcomes than TAU at post-treatment and at 9 months? Secondary question: Are effects larger for SCD than MCI? No medicines are used and risks are minimal. If effective, this scalable, low-cost, non-pharmacological approach could complement usual care for people in very early cognitive decline.

DETAILED DESCRIPTION:
Background Dementia affects tens of millions of people and no curative therapy exists. Non-pharmacological interventions that are safe, scalable, and acceptable are therefore essential to delay decline and preserve functioning. Positive Psychology Interventions (PPIs) have shown promising effects on wellbeing and, more recently, on cognitive performance and neural markers in older adults with early cognitive decline. Positive Neuropsychology proposes that cultivating positive traits and eudaimonic wellbeing may support brain plasticity and cognitive control through multiple pathways, including increased engagement, motivation, and adoption of protective lifestyles. Building on this framework, the present trial tests an online, multi-component PPI tailored for adults with Subjective Cognitive Decline (SCD) or Mild Cognitive Impairment (MCI). The program is designed to be feasible, scalable, and low-risk, and to generate clinically relevant outcomes on cognition and brain functioning.

Objectives and Hypotheses Primary objective: determine whether the PPI produces greater improvements than Treatment As Usual (TAU) in (a) cognitive performance and (b) neurophysiological indices of brain functioning at post-intervention and at 9-month follow-up. Secondary objectives: evaluate effects on wellbeing and related psychosocial constructs (character strengths, mindfulness), and assess feasibility, adherence, and safety of online delivery. We hypothesize larger gains with PPI at 16 weeks and sustained benefits at follow-up, with potentially stronger effects in SCD than MCI.

Study Design and Setting Randomized, parallel-group, superiority behavioral trial with two diagnostic groups (SCD, MCI) recruited via Alzheimer Hellas. Within each cohort, participants are randomized 1:1 to PPI or TAU, yielding four arms (SCD-PPI, SCD-TAU, MCI-PPI, MCI-TAU). Randomization is concealed and performed by site personnel who are not involved in outcome assessment. The trial is minimal risk, uses no FDA-regulated products, and is approved by the Bioethics Committee of Alzheimer Hellas (Approval No. 99/5-6-2024). Outcome assessors are trained and, where feasible, blinded to assignment.

Participants Community-dwelling older adults with a documented diagnosis of SCD or MCI from Alzheimer Hellas according to site procedures are eligibl. Key capabilities include informed consent, sufficient sensory ability for testing, and access/ability to join online groups. Major neurological/psychiatric conditions that would confound outcomes, severe sensory impairment preventing testing, and concurrent participation in similar psychological programs during the trial are excluded. After consent, participants receive unique study IDs; identifiers are stored separately, with controlled access, and destroyed after data lock.

Intervention: Multicomponent Positive Psychology Program Delivery: weekly small-group videoconference sessions (~60 minutes) for 16 weeks led by trained psychologists.

Assessment schedule and procedures

Assessments occur at four time points:

T0 baseline (pre-randomization); T1 mid-intervention (~6 weeks); T2 post-intervention (~16 weeks; primary endpoint); T3 follow-up (~9 months post-T2). Attendance and home-practice adherence are tracked. Adverse events (AEs) are monitored each visit and during sessions per institutional policy.

Outcomes and Data Acquisition

Primary outcomes (analyzed from T0 to T3):

Cognitive performance: a composite derived from the REMEDES4Alzheimer computerized battery capturing episodic memory, working memory, attention subdomains, and executive functions, with minimized demographic bias.

Brain functioning: EEG and functional near-infrared spectroscopy (fNIRS) markers obtained during standardized cognitive tasks using harmonized acquisition and artifact-handling protocols.

Secondary outcomes: validated indices of wellbeing (PERMA-Profiler; PANAS) measured at all time points to model trajectories. Exploratory psychosocial measures include character strengths (VIA-114GR) and mindfulness (MAAS). Feasibility metrics include recruitment and retention, session attendance, and self-reported practice.

Sample Size and Power Four arms (SCD-PPI, SCD-TAU, MCI-PPI, MCI-TAU). A priori power calculations indicate a minimum of 32 participants per arm; target enrollment N=128.

Data management and quality control Data are captured on secure, password-protected platforms under unique study IDs; personally identifying information is maintained in a separate, access-restricted file. Quality procedures include range and logic checks, double verification of key variables, and standardized preprocessing pipelines for EEG/fNIRS feature extraction. After database lock, the re-identification log is destroyed. De-identified data may be shared as described in the IPD plan.

Statistical analysis Analyses follow the intent-to-treat principle with participants analyzed as randomized. For longitudinal outcomes, linear mixed-effects models estimate change and Arm×Time interactions, with random intercepts for participants and adjustment for diagnosis cohort (SCD/MCI) and prespecified covariates (e.g., age, sex, baseline value). The two primary outcomes will be tested with appropriate multiplicity control. EEG/fNIRS features are derived via prespecified pipelines and analyzed analogously. Exploratory mediation models will assess whether changes in mindfulness or strengths use relate to cognitive and neural changes.

Safety and ethics Risks are minimal (time burden; potential fatigue during EEG and fNIRS). Standardized procedures and scheduled breaks mitigate burden. AEs are recorded, assessed for relatedness and severity, and reported to the ethics committee per policy. The study complies with the Declaration of Helsinki and applicable data-protection laws.

Implementation and expected impact Remote delivery enhances access for older adults with mobility or caregiving constraints and lowers cost for participants and providers. If efficacious, the program can be scaled across community and clinical settings through brief facilitator training and manualized materials. The trial will provide mechanistic evidence on whether cultivating character strengths and mindfulness improves cognitive functioning and alters neural activity in early decline. Demonstration of sustained benefits at nine months would support PPIs as practical, low-risk adjuncts to usual care for SCD and MCI, with potential to delay progression.

Follow-up and data sharing All participants are invited to T3 follow-up to assess durability. De-identified datasets may be shared on reasonable request after publication, subject to approvals and data-use agreements, consistent with the IPD sharing plan.

ELIGIBILITY:
Inclusion Criteria

-Documented diagnosis of Subjective Cognitive Decline (SCD) or Mild Cognitive Impairment (MCI) according to clinical evaluation and site standard criteria.

Exclusion Criteria

* Diagnosis of dementia (major neurocognitive disorder) or other major neurocognitive disorder that is moderate or severe.
* Major psychiatric disorder currently unstable or untreated (e.g., major depression with psychotic features, bipolar disorder, schizophrenia).
* Neurological conditions that affect cognition.
* Uncorrected hearing or vision problems that prevent participation in assessments or online sessions.
* Concurrent participation in another interventional study targeting cognition or wellbeing during the study period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Global cognitive composite (z-score) from REMEDES4Alzheimer | T0: Baseline prior to randomization T1: Mid-intervention at 6 weeks T2: Post-intervention at 16 weeks (primary endpoint) T3: Nine-month follow-up after T2
  Composite derived from REMEDES4Alzheimer subtests covering episodic memory, working memory, attention subdomains, and executive functions. Raw scores are standardized to z using baseline means,SDs and averaged to a global composite (higher scores indicate better cognition).
  Unit of measure: z-score (higher = better)
Resting-state fNIRS functional connectivity (HbO) between bilateral dorsolateral prefrontal cortices | T0 (Baseline), T2 (~16 weeks; primary endpoint), T3 (~9 months after T2) Unit of measure: Fisher z-transformed correlation coefficient (higher = stronger connectivity)
  Resting-state fNIRS recorded for 5-8 minutes (eyes-open fixation). Oxygenated hemoglobin (HbO) signals are preprocessed with motion-artifact correction, short-channel regression (if available), and band-pass filtering (e.g., 0.01-0.1 Hz). Functional connectivity is computed as the Pearson correlation between left and right DLPFC regions of interest and converted to Fisher z for analysis.
EEG alpha power at rest (eyes-closed) | Time Frame: T0 (Baseline), T2 (~16 weeks; primary endpoint), T3 (~9 months after T2)
  Mean absolute power in the 8-12 Hz band during 3-min resting eyes-closed, averaged across parieto-occipital electrodes; processed with artifact rejection and ICA according to prespecified pipeline.
  μV² (higher = better/according to hypothesis)

SECONDARY OUTCOMES:
Character Strengths total score (VIA-114GR) | T0: Baseline prior to randomization T1: Mid-intervention at 6 weeks T2: Post-intervention at 16 weeks (primary endpoint) T3: Nine-month follow-up after T2
  VIA-114GR total (or mean) score; subscales analyzed exploratorily. Unit of measure: total/mean score (higher = greater strengths use)
Wellbeing - PERMA-Profiler total score | T0: Baseline prior to randomization T1: Mid-intervention at 6 weeks T2: Post-intervention at 16 weeks (primary endpoint) T3: Nine-month follow-up after T2
  Total PERMA score; domain scores (P, E, R, M, A) examined secondarily. Unit of measure: score 0-10 (higher = better wellbeing)
Mindfulness (MAAS total) | T0: Baseline prior to randomization T1: Mid-intervention at 6 weeks T2: Post-intervention at 16 weeks (primary endpoint) T3: Nine-month follow-up after T2
  Mean of the Mindful Attention Awareness Scale. Unit of measure: mean score 1-6 (higher = greater mindfulness)
Positive Affect (PANAS) | T0 (Baseline), T2 (~16 weeks; primary endpoint), T3 (~9 months after T2)
  PANAS Positive Affect subscale. Negative Affect analyzed exploratorily. Unit of measure: score 10-50 (higher = more positive affect)

CONTACTS AND LOCATIONS:
Overall Officials: Despoina Moraitou, Professor, PhD, Principal Investigator — Aristotle University of Thessaloniki, Department of Psychology
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://doi.org/10.4236/psych.2021.123025
- See also: Related Info — https://doi.org/10.31234/osf.io/db3mk
- See also: Related Info — https://doi.org/10.5502/ijw.v6i3.526
- See also: Related Info — https://alzheimersnewstoday.com/mild-alzheimers-early-stage/
- See also: Related Info — https://doi.org/10.1016/j.chb.2009.02.003
- See also: Related Info — https://doi.org/10.1007/s12144-019-00236-7
- See also: Related Info — https://doi.org/10.1007/s10902-022-00598-z